CLINICAL TRIAL: NCT04087564
Title: Investigating Differences in Modulation of Nociceptive Processing by Music in Chronic Pain Patients
Brief Title: The Impact of Music on Nociceptive Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kristin Schreiber, Assistant Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019P000824
Record Dates: First submitted 2017-11-13; First posted 2019-09-12 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Pain, Acute; Pain, Chronic; Anxiety; Anxiety Disorders; Catastrophization; Healthy
Keywords: Music
MeSH Terms: conditions — Acute Pain; Chronic Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Each subject serves as their own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- music intervention (Experimental): Healthy volunteers, and patients diagnosed with HIV or fibromyalgia will complete 4 rounds of QST testing; baseline + 3 music conditions to determine effect of music on pain sensitivity.
  Interventions: Other: music intervention

INTERVENTIONS:
Other: music intervention — The music intervention (Unwind), developed by the investigators collaborators at the Sync Project, is a machine learning protocol that generates specific sounds and phrases of music that are stitched into a music track in response to user-reported pain, anxiety and catastrophizing scales. Unwind is delivered via a web application on a smart phone.
  Participants will also listen to white noise and their favorite music throughout the study session
  Other Names: Unwind; Favorite Music; White Noise

SUMMARY:
The investigators are studying the ways that different music may change pain perception

DETAILED DESCRIPTION:
In this study, the investigators are comparing healthy individuals to HIV and Fibromyalgia patients. The investigators are measuring the differences in pain processing between subject groups in the presence and absence of different music and distraction conditions. The investigators will be using Quantitative Sensory Testing (QST) in order to induce varying pain conditions on the participants. The investigators will also have participants complete sets of psychosocial questionnaires. Patients with Fibromyalgia tend to have a higher pain sensitivity. Additionally, patients with an HIV diagnosis tend to be prescribed opioid medications. The investigators would like to find out if music can modulate pain, and in turn help reduce the amount of opioid medications those with a chronic pain diagnosis take.

ELIGIBILITY:
Healthy volunteers no longer needed for this study (9/9/2021).

Inclusion criteria for Healthy volunteers (N=70) without a diagnosis of neuropathy or chronic pain:

* aged >18 years
* able to speak and understand English
* willingness to undergo psychophysical and psychosocial testing.

Exclusion criteria:

* diagnosed hearing loss
* diagnosis of chronic pain/neuropathy
* history of chronic opioid use (having an opioid prescription >30 days).

Inclusion criteria for Fibromyalgia patients: N=70:

* aged >18 years
* have a diagnosis of fibromyalgia with concurrent chronic pain for > 6 months, and meet the Wolfe et al 2011 research criteria for fibromyalgia
* have an average self-reported pain score of 4/10 or greater
* willing to undergo psychophysical and psychosocial testing
* able to speak and understand English.

Exclusion criteria:

--diagnosed hearing loss.

HIV Patients with chronic pain: N=70

* aged >18- years
* have a diagnosis of HIV infection
* have had chronic pain with onset > 6 months
* have an average self-reported pain score of 4/10 or greater
* willing to undergo psychophysical and psychosocial testing
* able speak and understand English.

Exclusion criteria:

--diagnosed hearing loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Modulation of Pressure Pain Threshold/Tolerance | 15 minutes
  Pressure algometry is the most commonly used test for static mechanical pressure sensation in the skin and in deep tissues. Pressure algometers deliver a firm and quantifiable pressure through a flat base applied to the skin. The electronic pressure algometer that we will use (Wagner Instruments) is a hand-held algometer utilizing a pressure-sensitive strain gauge, covered by a 0.5 cm2 circular probe. The probe is covered with a soft polypropylene disk, to avoid injury to the skin. The pressure applied through the probe is transduced, amplified, and converted to electrical reading on a digital display. The pressure will be slowly increased (1 lb/s) and the participant will be asked to note when they first feel pain and when they want the pressure to stop , which will be recorded as the pressure pain threshold and tolerance, respectively. This process will be repeated on the trapezius and the forearm, alternating between sides of the body with 20 seconds between measurements.
Modulation of Temporal Summation with Repeated Pinpricks | 15 minutes
  Will be assessed using standardized weighted pinprick applicators using a range of forces (128 mN, 256mN and 512mN) which result in a painful sensation in most subjects. First, a single stimulation of the lower force pinprick will be applied to the dorsal aspect of the index finger between the first and second interphalangeal joints of each hand while resting palm down on the armrest, and then rated by the subject on a scale of 0-10. The weight probe that induces at least some pain, but not more than 3/10 pain will be determined, and this probe used for repeated testing. Then, a train of 10 stimuli will be applied at the same spot, at a rate of 1 stimulation/second. The subject will rate pain on a scale of 0-10 after the first, fifth and tenth stimulus, then rate any ongoing pain 15 seconds after cessation of the last stimulus (painful after-sensations). Temporal summation will be calculated as the change in pain score between the highest and lowest pain ratings in a train.
Modulation of Temporal Summation with Pressure Cuff | 15 minutes
  Will be assessed through response to cuff pressure algometry (CPA), in a similar manner to our previous studies.123 Tonic, deep-tissue, mechanical stimulation will be applied using a rapid cuff inflator (Hokanson) wrapped around the leg, centered around the middle of the gastrocnemius muscle. Pressure will then be increased at approximately 5-10 mmHg/s, at which time participants will be asked to note when they first start feeling pain and then when they feel as though the pain is a 5/10. At this point the cuff will be deflated. Participants will be given a 30 second break. The cuff will be re-inflated to this previously identified pressure and held for two minutes (or until participant asks to stop), at which point the cuff will be deflated. Participants will be asked to rate their pain every 30 seconds, as well as to rate any painful after sensations. Temporal summation will be calculated as the change in pain score between the highest and lowest pain ratings in the 2 minutes.
Modulation of Heat Pain Threshold and Tolerance | 15 minutes
  Heat pain responses will be assessed using a contact thermode, which delivers heat stimuli through a computer-controlled system (Medoc). The contact probe will be positioned on the skin and affixed in place on the volar aspect of the non-dominant forearm with a soft Velcro strap, after which an ascending method of limits paradigm will be employed, using a rate of rise of 2°C/sec, starting at a baseline of 35°C. For heat pain threshold, subjects are instructed to press a button when the thermal stimulation first becomes painful; pressing the button returns the thermode temperature to 35°C. Then the thermode will again increase in temperature, and this time the conductor will ask the participant to press the button when the thermal stimulation reaches 5/10 pain, which will return the thermode temperature to 35°C.
Modulation of Heat Offset Analgesia | 15 minutes
  In order to measure offset analgesia the thermode will be ramped up to a temperature that is 1 degree less than the temperature that they indicated produced 5/10 pain. The temperature will be held for 5 seconds and the participant will be asked to provide a pain rating from 0-10 at the timepoint approximately 2 seconds into the 5 second period. Then the temperature will ramp up 1 degree higher (to the patient's 5/10 temperature) and held for 5 seconds. The participant will be asked to provide a pain rating from 0-10 at the timepoint approximately 2 seconds into the 5 second period. Then the temperature will return back to 1 degree lower, be held here for 5 seconds, and the participant will be asked to provide a pain rating from 0-10 at the timepoint approximately 2 seconds into the 5 second period. Lastly, the thermode will return to baseline temperature, and be removed from the forearm. The conductor will ask for pain scores every 7 seconds for 21 seconds seconds(aftersensations).
Modulation of Conditioned Pain Modulation | 15 minutes
  CPM will be measured by adaptations of testing procedures used in our previous studies.
  To measure CPM, pressure pain threshold and tolerance as measured earlier in the session will be compared to measurement in the presence of a conditioning stimulus (cold pain in hand). The participant will be asked to submerge their right hand (up to above the wrist) into a cold-water bath set at 6°C. Approximately 5 seconds after placing hand in cold water bath, a constant, increasing pressure (1lb/s) will again be applied to the contralateral trapezius with participant indicating when they start to feel pain (threshold) and when they want pressure to stop (tolerance). CPM defined as: CPM=((pressure pain in presence- pressure pain in absence of cold pain)/pressure pain in absence of cold pain)*100). Participants then asked to describe their worst cold pain, clinical pain, anxiety rating about testing and about the cold-water bath specifically, and if they experience any painful after sensations.
Modulation of Anxiety | 10 Minutes
  Question assessing how much anxiety felt during session, using Likert Scale (0-10), with 0 being no anxiety and 10 being extremely anxious.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Schreiber, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wilson JM, Franqueiro AR, Edwards RR, Chai PR, Schreiber KL. Individuals with fibromyalgia report greater pain sensitivity than healthy adults while listening to their favorite music: the contribution of negative affect. Pain Med. 2024 May 2;25(5):352-361. doi: 10.1093/pm/pnae005. PMID 38291916
- [Derived] Colebaugh CA, Wilson JM, Flowers KM, Overstreet D, Wang D, Edwards RR, Chai PR, Schreiber KL. The Impact of Varied Music Applications on Pain Perception and Situational Pain Catastrophizing. J Pain. 2023 Jul;24(7):1181-1192. doi: 10.1016/j.jpain.2023.01.006. Epub 2023 Jan 14. PMID 36646399